CLINICAL TRIAL: NCT03530267
Title: Aflibercept and 5-FU vs. FOLFOX as 1st Line Treatment for Elderly or Frail Elderly Patients With Metastatic Colorectal Cancer
Brief Title: Aflibercept and 5-FU vs. FOLFOX as 1st Line Treatment for Elderly or Frail Elderly Patients With Met. Colorectal Cancer
Acronym: ELDERLY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Collaborators: STABIL - Statistische und Biometrische Lösungen (Unknown); Trium Analysis Online GmbH (Industry); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ELDERLY
Record Dates: First submitted 2018-05-08; First posted 2018-05-21 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; 5-FU; Aflibercept; Oxaliplatin
MeSH Terms: conditions — Colorectal Neoplasms | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (mFOLFOX7) (Active Comparator): Patients in the 5-FU / oxaliplatin arm receive modified (m) FOLFOX 7: Folinic acid 350 mg/m² and oxaliplatin 68 mg/m² by concurrent 2-h intravenous infusion, 5-fluorouracil 1920 mg/m² 46-h intravenous infusion every 2 weeks (qd15).
  This regimen represents the 80% dosage reduced mFOLFOX 7. The 80% dose reduction was shown to be a tolerable regimen in frail elderly patients in the FOCUS 2 study.
  Interventions: Drug: mFOLFOX7
- Arm B (Aflibercept + mLV5FU2) (Experimental): Patients in the 5-FU / aflibercept arm receive aflibercept 4mg/kg as 1-h infusion followed by folinic acid 350 mg/m² by 2-h intravenous infusion, 5-fluorouracil 1920 mg/m² 46-h intravenous infusion (mLV5FU2) every 2 weeks (qd15).
  The decision to use reduced doses of 5-FU and folinic acid was made to have comparable doses to the reduced FOLFOX 7.
  Interventions: Drug: Aflibercept + mLV5FU2

INTERVENTIONS:
Drug: Aflibercept + mLV5FU2 — Patients receive aflibercept 4mg/kg as 1-h infusion followed by folinic acid 350 mg/m² by 2-h intravenous infusion, 5-fluorouracil 1920 mg/m² 46-h intravenous infusion (mLV5FU2) every 2 weeks (qd15).
  Arms: Arm B (Aflibercept + mLV5FU2)
Drug: mFOLFOX7 — Patients in this arm receive modified (m) FOLFOX 7: Folinic acid 350 mg/m² and oxaliplatin 68 mg/m² by concurrent 2-h intravenous infusion, 5-FU 1920 mg/m² 46-h intravenous infusion every 2 weeks (qd15).
  Arms: Arm A (mFOLFOX7)

SUMMARY:
This is a controlled, open-label, randomized phase- II trial (1:1 randomization) investigating 5-FU + aflibercept and 5-FU + oxaliplatin in elderly and frail elderly patients with mCRC scheduled to receive first line treatment.

DETAILED DESCRIPTION:
The current trial seeks to evaluate a new treatment option for elderly / frail elderly patients with mCRC including 5-FU - better tolerated than capecitabine in the FOCUS2 study - in conjunction with aflibercept, a broad active anti-angiogenic drug within a randomized phase-II setting. Patients will be randomized using a 1:1 randomization between 5-FU / aflibercept and 5-FU / oxaliplatin using the oxaliplatin-based regimen established in FOCUS2 trial. Main goal is to estimate the 6-months PFS rate with 5-FU / Aflibercept and the safety of this regimen. The decision to use a randomized phase-II design using the "FOCUS2- FOLFOX" is based on two assumptions; (i) Bias can be better controlled by using a randomized phase-II design (ii) A clear standard regimen in frail elderly cannot be defined, but FOLFOX was superior to 5-FU alone in FOCUS2 and the patient population included in the FOCUS2 study represents the patient population scheduled to be included in the current trial.

Provided the randomized phase-II study shows adequate efficacy of 5-FU / aflibercept and a tolerable safety profile, the study will be carried on to the phase-III part of the trial. Description of the terms and conditions to expand the current trial are not part of this protocol. Briefly, a potential phase-III study should aim at showing non-inferiority of 5-FU / aflibercept regarding 6-months PFS rate as primary endpoint. This would allow to include all patients from the phase-II part in the phase-III study in order to save time and patients.

ELIGIBILITY:
Inclusion Criteria:

1. To enter this trial the oncologist has to confirm, that the patient was in his or her opinion not a candidate for standard full-dose combination therapy. Moreover, the oncologist has to state the reason for entering the trial (Advanced age alone versus both age and frailty). As an operational definition for frailty the G8 screening tool will be used upon inclusion of the patient in a standardized manner. Briefly, G8 is an established screening tool that includes seven items from the Mini Nutritional Assessment (MNA) and an age-related item (<80, 80 to 85, or 85 years). The total score can range from 0 to 17. The result on the G8 is considered abnormal if the score is ≤14, indicating a geriatric risk profile.
2. Patients have to have histologically confirmed mCRC with unidimensionally measurable inoperable advanced or metastatic disease
3. ECOG performance status of 2 or better.
4. Life expectancy of 3 months or longer at enrolment
5. Patients >70 years with no upper age limit
6. Previous adjuvant chemotherapy is allowed if completed more than 6 months before randomisation
7. Previous rectal (chemo)radiotherapy is allowed if completed more than 6 months before randomisation
8. Hematological status:

   * Neutrophils (ANC) ≥ 1.5 x 109/L
   * Platelets ≥ 100 x 109/L
   * Hemoglobin ≥ 9 g/dL
9. Adequate renal function:

   • Serum creatinine level ≤ 1.5 x upper limit normal (ULN)
10. Adequate liver function:

    * Serum bilirubin ≤ 1.5 x upper limit normal (ULN)
    * Alkaline phosphatase ≤ 2.5 x ULN (unless liver metastases are present, then < 5 x ULN in that case)
    * AST and ALT < 3 x ULN (unless liver metastases are present then < 5 x ULN in that case)
11. Proteinuria < 2+ (dipstick urinalysis) or ≤ 1 g/24hour
12. Signed and dated informed consent, and willing and able to comply with protocol requirements
13. Regular follow-up feasible
14. Male patients with a partner of childbearing potential must agree to use effective contraception (Pearl Index < 1) during the course of the trial and at least 3 months after last administration of the study drug.

Exclusion Criteria:

1. Prior systemic chemotherapy for mCRC
2. Other concomitant or previous malignancy, except:

   * Adequately treated in-situ carcinoma of the uterine cervix
   * Basal or squamous cell carcinoma of the skin
   * Cancer in complete remission for > 5 years
3. Any other serious and uncontrolled non-malignant disease, major surgery or traumatic injury within the last 28 Days
4. History or evidence upon physical examination of CNS metastasis unless adequately treated (irradiation and no seizure with appropriate treatment)
5. Uncontrolled hypercalcemia
6. Pre-existing peripheral neuropathy (NCI grade ≥2)
7. Concomitant protocol unplanned antitumor therapy (e.g. chemotherapy, molecular targeted therapy, immunotherapy),
8. Treatment with any other investigational medicinal product within 28 days prior to study entry.
9. Significant cardiovascular disease:

   * Cardiovascular accident or myocardial infarction or unstable angina ≤6 months before start of study treatment
   * Severe cardiac arrhythmia
   * New York Heart Association grade ≥2 congestive heart failure
   * Uncontrolled hypertension (defined as systolic blood pressure >150 mmHg and/or diastolic blood pressure >100 mmHg), or history of hypertensive crisis, or hypertensive encephalopathy.
   * History of stroke or transient ischemic attack ≤6 months before start of study treatment
   * Coronary/peripheral artery bypass graft ≤6 months before start of study treatment.
   * Deep vein thrombosis or thromboembolic events ≤1 month before start of study treatment
10. Patients with known allergy to any excipient to study drugs,
11. Any of the following within 3 months prior to randomization: Grade 3-4 gastrointestinal bleeding/hemorrhage, treatment resistant peptic ulcer disease, erosive oesophagitis or gastritis, infectious or inflammatory bowel disease, diverticulitis, pulmonary embolism or other uncontrolled thromboembolic event.
12. Bowel obstruction.
13. Treatment with CYP3A4 inducers unless discontinued > 7 days prior to randomization
14. Known dihydropyrimidine dehydrogenase (DPD) deficiency
15. Involvement in the planning and/or conduct of the study (applies to both Sanofi staff and/or staff of sponsor and study site)
16. Patient who might be dependent on the sponsor, site or the investigator
17. Patient who has been incarcerated or involuntarily institutionalized by court order or by the authorities § 40 Abs. 1 S. 3 Nr. 4 AMG.
18. Patients who are unable to consent because they do not understand the nature, significance and implications of the clinical trial and therefore cannot form a rational intention in the light of the facts [§ 40 Abs. 1 S. 3 Nr. 3a AMG].

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 124 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 6 months
  Rate of patients free of progression

SECONDARY OUTCOMES:
Safety: Dose intensities of study medication | 6 months
  As calculated over the whole treatment duration and summarized descriptively by summary statistics.
Safety: Adverse events (AE) | 7 months
  AE's will be summarized by presenting the number and percentages of patients having any AE
Safety: Dose modification of study drug due to adverse events | 6 months
  Dose modifications, including discontinuations, will be summarized by presenting the number and percentages of patients having any dose modification
Safety: Rate of treatment discontinuation due to toxicitiy | 6 months
  Rate of treatment discontinuations during the study
Safety: Laboratory abnormalities | 6 months
  Summary of lab abnormalities as assessed in the documentation
Efficacy: Response rates | 2 years
  As measured by RECIST criteria v. 1.1
Efficacy: Overall survival (OS) | 2 years
  OS according to Kaplan-Meier
Efficacy: PFS | 2 years
  PFS according to Kaplan-Meier
Patient reported outcomes (PRO): Quality of life | 6 months
  Quality of life (QoL) as measured by EQ-5D-5L at d1 of each cycle and on EOT.
PRO: Geriatric assessment | 6 months
  Geriatric assessment as measured by using G8, ADL and IADL
PRO: Overall treatment utility | 6 months
  Overall treatment utility is evaluated according to the principles used in the FOCUS2 trial. Cf. Seymour et al. Geriatric oncol 2013.

CONTACTS AND LOCATIONS:
Overall Officials: Salah-Eddin Al-Batran, Prof. Dr., Study Chair — Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest
Locations (25):
- Germany (25):
  - Phase Drei, Aschaffenburg
  - HELIOS Klinikum Bad Saarow, Bad Saarow
  - Klinikum Bayreuth, Bayreuth
  - MVZ Seestrasse, Berlin
  - Klinikum Bremen Nord, Bremen
  - Kliniken Essen-Mitte, Essen
  - Agaplesion Markus Krankenhaus, Frankfurt
  - Krankenhaus Nordwest GmbH, Frankfurt
  - Klinikum Garmisch-Partenkirchen GmbH, Garmisch-Partenkirchen
  - Nationales Centrum für Tumorerkrankungen (NCT), Heidelberg
  - Städtisches Klinikum Karlsruhe, Karlsruhe
  - DRK-Kliniken Nordhessen gGmbH, Kassel
  - Ortenau Klinikum Lahr, Lahr
  - Onkologisches Zentrum, Lebach
  - Klinikum Ludwigshafen, Ludwigshafen
  - Klinikum Magdeburg gGmbH, Magdeburg
  - Tagestherapiezentrum am ITM Universitätsmedizin Mannheim, Mannheim
  - Kliniken Ostalb, Mutlangen
  - Klinikum der Universität München-Großhadern, München
  - Kliniken des Landkreises Neumarkt in der Oberpfalz, Neumarkt in der Oberpfalz
  - Studienzentrum Onkologie Ravensburg, Ravensburg
  - Clinical Research Stolberg GmbH, Stolberg
  - Klinikum Mutterhaus Trier, Trier
  - Universitätsklinikum Tübingen, Tübingen
  - Klinikum Wilhelmshaven, Wilhelmshaven

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared

REFERENCES:
- [Background] Seymour MT, Thompson LC, Wasan HS, Middleton G, Brewster AE, Shepherd SF, O'Mahony MS, Maughan TS, Parmar M, Langley RE; FOCUS2 Investigators; National Cancer Research Institute Colorectal Cancer Clinical Studies Group. Chemotherapy options in elderly and frail patients with metastatic colorectal cancer (MRC FOCUS2): an open-label, randomised factorial trial. Lancet. 2011 May 21;377(9779):1749-59. doi: 10.1016/S0140-6736(11)60399-1. Epub 2011 May 11. PMID 21570111